CLINICAL TRIAL: NCT00723957
Title: A Randomized Phase 2 Study of Ixabepilone Plus Carboplatin and Paclitaxel Plus Carboplatin in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: A Randomized Phase 2 Study of Ixabepilone Plus Carboplatin and Paclitaxel Plus Carboplatin in Advanced Nonsmall-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-163
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Advanced/Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ixabepilone; Paclitaxel; BMS 181339; Carboplatin; Area Under Curve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) (Experimental)
  Interventions: Drug: Ixabepilone, 32 mg/m^2; Drug: Carboplatin (area under the concentration curve [AUC] 6)
- Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6) (Active Comparator)
  Interventions: Drug: Paclitaxel, 200 mg/m^2; Drug: Carboplatin (area under the concentration curve [AUC] 6)

INTERVENTIONS:
Drug: Ixabepilone, 32 mg/m^2 — Intravenous (IV) solutions, ixabepilone, 32 mg/m^2
  Other Names: IXEMPRA; BMS-247550
  Arms: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6)
Drug: Paclitaxel, 200 mg/m^2 — IV solutions, paclitaxel, 200 mg/m^2
  Other Names: TAXOL; BMS-181339; PARAPLATIN; BMY-26575
  Arms: Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Drug: Carboplatin (area under the concentration curve [AUC] 6) — Carboplatin (AUC 6) day 1, every 21 days, 6 cycles

SUMMARY:
The purpose of this study is to determine whether progression-free survival with ixabepilone is superior to that achieved with paclitaxel plus carboplatin in participants with advanced nonsmall-cell lung cancer and beta III (βIII)-tubulin-positive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC)(squamous cell, adenocarcinoma, large cell, or bronchoalveolar carcinoma)
* Stage IIIB NSCLC with pleural effusion, Stage IV NSCLC, or recurrent disease following surgery with or without radiation therapy
* Available paraffin-embedded tissue to measure the expression levels of βIII tubulin
* Disease measurable by Response Evaluation Criteria in Solid Tumors, with at least 1 target lesion situated outside any previous radiotherapy field
* Karnofsky performance status of 70-100
* Life expectancy of at least 3 months
* Men and women, ages 18 years and older

Exclusion Criteria:

* Uncontrolled brain metastases
* Peripheral neuropathy greater than Grade 1
* Fewer than 4 weeks from prior radiation therapy or locoregional surgeries to randomization date (less than 1 week from focal/palliative radiotherapy or minor surgery)
* Any concurrent malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix
* Known HIV-positive status
* Absolute neutrophil count lower than 1500 cells mm^3
* Total bilirubin level higher than upper limit of normal (ULN) as defined by the institution (with the exception of elevation due to Gilbert's syndrome)
* Aspartate transaminase or alanine transaminase level higher than 2.5*ULN
* Serum creatine level of 1.5 mg/dL or higher
* Renal function with a creatinine clearance of less than 50 mL/min (as calculated with the Cockcroft and Gault equation)
* Any prior antineoplastic systemic regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (2):
  - Scripps Cancer Center, La Jolla, California
  - Uof Md,Greenebaum Cancer Ctr., Baltimore, Maryland
- Argentina (2):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Buenos Aires
- Australia (3):
  - Local Institution, Bankstown, New South Wales
  - Local Institution, Frankston, Victoria
  - Local Institution, Nedlands, Western Australia
- France (2):
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (3):
  - Local Institution, Bad Berka
  - Local Institution, Großhansdorf
  - Local Institution, Ulm
- Italy (4):
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Sondrio
  - Local Institution, Terni
- Russia (5):
  - Local Institution, Chelyabinsk
  - Local Institution, Kazan'
  - Local Institution, Moscow
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
- South Korea (2):
  - Local Institution, Goyang-si, Gyeonggi-do
  - Local Institution, Seoul
- Local Institution, Baracaldo (Vizcaya), Spain
- Taiwan (3):
  - Local Institution, Taichung
  - Local Institution, Taipei
  - Local Institution, Taoyuan Hsien

REFERENCES:
- [Derived] Edelman MJ, Schneider CP, Tsai CM, Kim HT, Quoix E, Luft AV, Kaleta R, Mukhopadhyay P, Trifan OC, Whitaker L, Reck M. Randomized phase II study of ixabepilone or paclitaxel plus carboplatin in patients with non-small-cell lung cancer prospectively stratified by beta-3 tubulin status. J Clin Oncol. 2013 Jun 1;31(16):1990-6. doi: 10.1200/JCO.2012.45.3282. Epub 2013 Apr 15. PMID 23589560
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 260 participants enrolled, 197 were randomized. Among those randomized, 191 received treatment.
Groups:
- Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6): Ixabepilone administered as a 3-hour intravenous (IV) infusion at a starting dose of 32 mg/m^2 on Day 1 of a 21-day cycle followed by carboplatin, administered at a dose calculated to produce an area under the concentration-time curve (AUC) of 6 mg/mL per minute (AUC 6), on Day 1 of a 21-day cycle for a maximum of 6 cycles
- Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6): Paclitaxel administered as a 3-hour IV infusion at a starting dose of 200 mg/m^2 on Day 1 of a 21-day cycle followed by carboplatin, administered at a dose calculated to produce an AUC 6, on Day 1 of a 21-day cycle for a maximum of 6 cycles
Period: Overall Study
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Started | 98 (Randomized) | 99 (Randomized)
Completed | 47 (Completed 6 cycles of study drug (maximum per protocol)) | 46 (Completed 6 cycles of study drug (maximum per protocol))
Not Completed | 51 | 53
Not completed — Adverse event unrelated to study drug | 1 | 4
Not completed — Death | 3 | 4
Not completed — Disease progression | 27 | 25
Not completed — Maximum clinical benefit | 4 | 5
Not completed — Investigator decision | 1 | 1
Not completed — Study drug toxicity | 4 | 6
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Reason not analyzed | 1 | 0
Not completed — Never received treatment | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6) | Total
Number analyzed (Participants) | 98 | 99 | 197
Age, Customized [Median (Full Range); unit: Years] — Participants with beta III (βIII)-tubulin positive tumors
  Years
    Beta III (βIII)-tubulin positive tumors (n=53, 51) | 60.0 [29.0 to 80.0] | 60.0 [43.0 to 80.0] | 60.0 [29.0 to 80.0]
    βIII-tubulin negative tumors (N=45, 48) | 60.0 [35.0 to 78.0] | 60.5 [34.0 to 85.0] | 60.0 [34.0 to 85.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 67 | 139
  Male | 26 | 32 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 30 | 22 | 52
  White | 68 | 76 | 144
  Other | 0 | 1 | 1
Number of participants with βIII-tubulin positive and negative tumors [Number; unit: Participants]
  βIII tubulin-positive tumors | 53 | 51 | 104
  βIII tubulin-negative tumors | 45 | 48 | 93

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival in the Subgroup of Participants With βIII-tubulin Positive Tumors
Description: Progression-free survival is defined as the period from date of randomization to date of disease progression or death. For participants who do not progress or die at the end of the study, progression-free survival was censored at the last tumor assessment date. For those who have no on-study tumor assessment, progression-free survival was censored at the date of randomization. A tumor was considered to be beta III (βIII)-tubulin positive if 50% or more of the tumor cells had a βIII-tubulin immunohistochemistry staining intensity equal to or greater than that of the positive control.
Time Frame: Randomization to disease progression or death (maximum reached: 14.39 months )
Population: All randomized participants with βIII-tubulin positive tumors and who received study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 53 | 51
Months | 4.27 (NA) [2.89 to 5.65] | 4.27 (NA) [3.61 to 6.05]
Statistical Analysis 1: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.04, 90% CI 1-sided [upper limit 1.41]
Statistical Analysis 2: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); P-value is 1-sided; Test type: Superiority or Other; p = 0.5735, Log Rank

2. Secondary Outcome: Progression-free Survival in the Subgroup of Participants With βIII-tubulin Negative Tumors
Description: Progression-free survival is defined as the period from date of randomization to date of disease progression or death. For participants who do not progress or die at the end of the study, progression-free survival was censored at the last tumor assessment date. For those who have no on study tumor assessment, progression-free survival was censored at the date of randomization.
Time Frame: Randomization to disease progression or death (maximum reached: 12.29 months)
Population: All randomized participants who had βIII-tubulin positive tumors and who received study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 45 | 48
Months | 5.78 (NA) [5.29 to 8.41] | 5.32 (NA) [4.27 to 5.98]
Statistical Analysis 1: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.78, 90% CI 1-sided [upper limit 1.10]
Statistical Analysis 2: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); P-value is 1-sided; Test type: Superiority or Other; p = 0.1750, Log Rank

3. Secondary Outcome: Progression-free Survival in the Overall Population
Description: as for outcome 2
Time Frame: Randomization to disease progression or death, assessed to 12.29 months
Population: All randomized participants who received study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 98 | 99
Months | 5.29 [4.14 to 5.88] | 5.13 [4.21 to 5.78]
Statistical Analysis 1: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.92, 90% CI 1-sided [upper limit 1.15]
Statistical Analysis 2: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); P-value is 1-sided; Test type: Superiority or Other; p = 0.316, Log Rank

4. Secondary Outcome: Percentage of Participants With Best Response of Complete Response (CR) or Partial Response (PR)
Description: Response evaluated per Response Evaluaton in Solid Tumor (V1.0) guidelines and assessed using magnetic resonance imaging. Percentage of best response=the total number of participants with the best overall response of CR or PR divided by the total number of randomized participants in that treatment arm. CR=disappearance of all target lesions; PR=at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: At randomization and then every 6 weeks to date of CR, PR, or progression for 6 21-day cycles
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 98 | 99
Percentage of participants
  βIII-tubulin positive subgroup (n=53, n=51) | 17.0 [8.1 to 29.80] | 29.4 [17.5 to 43.8]
  βIII-tubulin negative subgroup (n=45, n=48) | 26.7 [14.6 to 41.9] | 27.1 [15.3 to 41.8]
  Overall population | 21.4 [13.8 to 30.9] | 28.3 [19.7 to 38.2]

5. Secondary Outcome: Time to Response
Description: Time to Response is defined as the time from randomization date until the date of first response (Partial Response [PR] or Complete Response [CR])
Time Frame: Randomization to date of first response (PR or CR)
Population: All randomized participants
Measure: Median (Full Range); unit: Weeks
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 21 | 28
Weeks
  Beta III positive (n=9, 15) | 12.1 [5.1 to 19.3] | 6.6 [5.3 to 18.1]
  Beta III negative (n=12, 13) | 9.5 [5.0 to 17.4] | 7.0 [5.1 to 12.9]
  Overall population | 12.1 [5.0 to 19.3] | 6.6 [5.1 to 18.1]

6. Secondary Outcome: Number of Participants With Death as Outcome, Drug-related Adverse Events (AEs), Serious AEs (SAEs), Drug-related SAEs, AEs Leading to Discontinuation, and Drug-related Peripheral Neuropathy
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related is defined as possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: Days 1 through 21, continuously
Population: All participants who received any investigational product.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 96 | 95
Participants
  Death | 28 | 34
  Drug-related AEs | 85 | 87
  SAEs | 27 | 28
  Drug-related SAEs | 15 | 9
  AEs Leading to Discontinuation | 11 | 15
  Drug-related peripheral neuropathy | 35 | 54

7. Secondary Outcome: Number of Participants With Hematology Laboratory Results of Grade 3 or 4
Description: LLN=lower level of normal. Leukocytes (leukopenia) Grade 1: <LLN to 3.0*10^9/L, Grade 2:<3.0 to 2.0*10^9/L, Grade 3: <2.0 to 1.0*10^9/L, Grade 4: <1.0*10^9/L; Neutrophils (neutropenia) Grade 1: <LLN to 1.5*10^9/L, Grade 2: <1.5 to 1.0*10^9/L, Grade 3: <1.0 to 0.5*10^9/L, Grade 4: <0.5*10^9/L; Platelet count(thrombocytopenia) Grade 1: LLN to 75.0*10^9/L, Grade 2: <75.0 to 50.0*10^9/L, Grade 3: <50.0 to 25.0*10^9/L, Grade 4:<25.0 to 10^9/L; Hemoglobin (anemia) Grade 1: <LLN to 10.0 g/dL, Grade 2: <10.0 to 8.0 g/dL, Grade 3: <8.0 to 6.5 g/dL, Grade 4: <6.5 g/dL.
Time Frame: At screening and weekly during 21-day cycle
Population: All participants who received any investigational product.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 96 | 95
Participants
  Leukopenia, Grade 3 or 4 | 31 | 15
  Neutropenia, Grade 3 or 4 | 54 | 51
  Thrombocytopenia, Grade 3 or 4 | 14 | 1
  Anemia, Grade 3 or 4 | 15 | 0

8. Secondary Outcome: Number of Participants With Grade 3 or 4 Abnormalities in Liver Function and Urine Laboratory Test Results
Description: ULN=upper level of normal. Alkaline phosphatase (ALP) Gr 1:>ULN to 2.5*ULN, Gr 2: >2.5 to 5.0*ULN, Gr 3: >5.0 to 20.0*ULN, Gr 4: >20.0*ULN; Aspartate aminotransferase (AST) Gr 1: >ULN to 2.5*ULN, Gr 2: >2.5 to 5.0*ULN, Gr 3: >5.0 to 20.0*ULN, Gr 4: >20.0*ULN
Time Frame: At screening and within 72 hours of start of 21-day cycle (Cycle 2 and beyond)
Population: All participants who received any investigational product.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 96 | 95
Participants
  ALP, Grade 3 | 1 | 0
  ALP. Grade 4 | 0 | 0
  AST, Grade 3 | 0 | 1
  AST, Grade 4 | 0 | 0

9. Secondary Outcome: Median Length of Survival in the Overall Population and in the Subgroups of Patients With βIII-tubulin Positive (β3T+) and βIII-tubulin Negative (β3T-)Tumors
Description: Overall Survival was computed for all randomized participants and was defined as the time between randomization and death. Participants who did not die at the end of the study were censored at their last known alive date.
Time Frame: Randomization to death or last known alive date, up to 31.34 months
Population: All participants randomized to receive treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Number analyzed (Participants) | 98 | 99
Months
  βIII-tubulin positive subgroup (n=53, 51) | 10.61 (NA) [7.16 to 13.96] | 11.37 (NA) [8.15 to 15.41]
  βIII-tubulin negative subgroup (n=45, 48) | 16.92 (NA) [13.04 to 27.96] | 9.40 (NA) [7.98 to 13.40]
  Overall population | 13.04 (NA) [9.99 to 14.52] | 10.15 (NA) [8.28 to 13.40]
Statistical Analysis 1: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.6, 90% CI 1-sided [upper limit 2.10] — β3T+ subgroup
Statistical Analysis 2: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.70, 90% CI 1-sided [upper limit 0.90] — β3T- subgroup
Statistical Analysis 3: Comparison: Ixabepilone, 32 mg/m^2 + Carboplatin (AUC 6) vs Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6); Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.10, 90% CI 1-sided [upper limit 1.40] — Overall population

ADVERSE EVENTS:
Groups:
- Ixabepilone, 32 mg/m^2 + Carboplatin (AUC): Ixabepilone administered as a 3-hour intravenous (IV) infusion at a starting dose of 32 mg/m^2 on Day 1 of a 21-day cycle followed by carboplatin, administered at a dose calculated to produce an area under the concentration-time curve (AUC) of 6 mg/mL per minute (AUC 6), on Day 1 of a 21-day cycle for a maximum of 6 cycles
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6)
Serious Adverse Events (participants affected / at risk) | 27/95 | 28/96
Other Adverse Events (participants affected / at risk) | 88/95 | 91/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC) (N=95) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6) (N=96)
BLOOD CREATININE INCREASED (Investigations) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 2 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 0
PERICARDITIS CONSTRICTIVE (Cardiac disorders) | 1 | 0
PHLEBITIS (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 2 | 1
HEADACHE (Nervous system disorders) | 1 | 0
MYELITIS (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 3 | 0
CONVULSION (Nervous system disorders) | 1 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 2
NAUSEA (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 3
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 4 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 3
FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHIAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OESOPHAGOBRONCHIAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PAIN (General disorders) | 0 | 1
FATIGUE (General disorders) | 1 | 1
PYREXIA (General disorders) | 1 | 2
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 2
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 32 mg/m^2 + Carboplatin (AUC) (N=95) | Paclitaxel, 200 mg/m^2 + Carboplatin (AUC 6) (N=96)
INSOMNIA (Psychiatric disorders) | 7 | 7
HYPERSENSITIVITY (Immune system disorders) | 2 | 6
HEADACHE (Nervous system disorders) | 5 | 7
DIZZINESS (Nervous system disorders) | 8 | 7
DYSGEUSIA (Nervous system disorders) | 4 | 6
PARAESTHESIA (Nervous system disorders) | 9 | 9
NEUROPATHY PERIPHERAL (Nervous system disorders) | 17 | 22
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 8 | 21
NAUSEA (Gastrointestinal disorders) | 41 | 31
VOMITING (Gastrointestinal disorders) | 17 | 10
DIARRHOEA (Gastrointestinal disorders) | 15 | 16
CONSTIPATION (Gastrointestinal disorders) | 12 | 13
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 6
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 30 | 27
ANAEMIA (Blood and lymphatic system disorders) | 25 | 13
LEUKOPENIA (Blood and lymphatic system disorders) | 12 | 10
NEUTROPENIA (Blood and lymphatic system disorders) | 32 | 22
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 17 | 1
RASH (Skin and subcutaneous tissue disorders) | 5 | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 45 | 55
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 9
MYALGIA (Musculoskeletal and connective tissue disorders) | 15 | 29
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 | 25
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 15
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 9
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 11 | 5
PAIN (General disorders) | 6 | 4
FATIGUE (General disorders) | 32 | 30
PYREXIA (General disorders) | 10 | 6
ASTHENIA (General disorders) | 12 | 17
CHEST PAIN (General disorders) | 10 | 14
OEDEMA PERIPHERAL (General disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.